CLINICAL TRIAL: NCT04840199
Title: Randomized, Controlled Trial to Evaluate the Anti-inflammatory Efficacy of Letermovir (Prevymis) in Adults With Human Immunodeficiency Virus (HIV)-1 and Asymptomatic Cytomegalovirus (CMV) Who Are on Suppressive ART and Its Effect on Chronic Inflammation, HIV Persistence, and Other Clinical Outcomes
Brief Title: A Study to Evaluate the Anti-inflammatory Effects of Letermovir (Prevymis) in Adults With Human Immunodeficiency Virus (HIV)-1 and Asymptomatic Cytomegalovirus (CMV) Who Are on Suppressive Antiretroviral Therapy, Plus Its Effect on Chronic Inflammation, HIV Persistence and Other Clinical Outcomes.
Acronym: ELICIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently closed to screening and accrual due to futility
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A5383; 38597 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: HIV Infections; Cytomegalovirus; CMV
MeSH Terms: conditions — HIV Infections | interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letermovir (Experimental): Participants randomized to letermovir for 48 weeks followed by 12 weeks off letermovir
  Interventions: Drug: Letermovir Oral Tablet
- No anti-CMV treatment (No Intervention): Participants randomized to no study intervention for 60 weeks

INTERVENTIONS:
Drug: Letermovir Oral Tablet — 480 mg administered orally once daily with or without food
  Other Names: Prevymis
  Arms: Letermovir

SUMMARY:
This was an open-label, controlled study, conducted at US sites to evaluate the anti-inflammatory effectiveness of the study drug letermovir in adults with HIV and asymptomatic cytomegalovirus (CMV) who were on antiretroviral therapy (ART)-mediated suppression. Participants were randomly assigned to receive either letermovir once daily or no anti-CMV treatment, for 48 weeks.

The primary hypothesis of this study was that letermovir would cause a greater reduction in plasma soluble receptor for tumor necrosis factor type II (sTNFRII) levels than no anti-CMV treatment at weeks 46/48.

DETAILED DESCRIPTION:
This was a phase 2, randomized, open-label, controlled, multicenter trial to evaluate the anti-inflammatory efficacy of letermovir, administered once daily for 48 weeks in adults with HIV and asymptomatic CMV, who are on ART-mediated suppression. Participants were randomized 1:1 to receive either letermovir or no anti-CMV treatment. The target enrollment was 180 participants.

A futility analysis was planned to be performed after the first 40 participants to initiate study treatment reached their 8-week study visit. Study enrollment was to be paused after the 40th participant started the study until the results of the futility analysis were considered.

This study was terminated due to futility.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

   * NOTE: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies.

   WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. More information on this criterion can be found in the protocol.
2. Currently on continuous combination ART (antiretroviral therapy) for ≥48 weeks prior to study entry. This is defined as continuous ART for the 48-week period prior to study entry with no ART interruption longer than 7 consecutive days.
3. Screening plasma HIV-1 RNA <40 copies/mL within 90 days prior to study entry using a FDA-approved assay with a quantification limit of 40 copies/mL or lower performed by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
4. HIV-1 RNA level <40 copies/mL for at least 48 weeks prior to study entry performed by any US laboratory that has a CLIA certification or its equivalent.

   * NOTE: Single determinations that are between the assay quantification limit and 500 copies/mL (i.e., "blips") are allowed as long as the preceding and subsequent determinations are below the level of quantification. The screening value may serve as the subsequent undetectable value following a blip.
5. CD4⁺/CD8⁺ cell count obtained within 90 days prior to study entry at any US laboratory that has a CLIA certification or its equivalent.
6. Positive CMV IgG serology, at any time prior to study entry using a FDA-approved assay at any US laboratory that has a CLIA certification or its equivalent.

   * NOTE: If a prior positive CMV IgG serology test is confirmed in the medical record, a repeat CMV IgG test is not required at screening.
7. The following laboratory values obtained within 90 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent:

   * Hemoglobin >9.0 g/dL
   * Platelet count >75,000/mm³
   * Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase ≤3 x ULN (upper limit of normal)
   * Total bilirubin ≤2.5 x ULN

     * NOTE: If an individual is taking atazanavir-containing regimen at the time of screening, a total bilirubin of ≤5 x ULN is acceptable.
   * Estimated Glomerular Filtration Rate (eGFR) >30 mL/min/1.73m² or creatinine clearance (CrCl) >30 mL/min using the Cockcroft-Gault, EPI-GFR or MDRD equations located on the DMC website.
8. For individuals assigned female sex at birth and of reproductive potential, negative serum or urine pregnancy test within 24 hours prior to study entry by any US clinic or laboratory that has a CLIA certification or its equivalent, or a CLIA Certificate of Waiver for those performing a point of care (POC)/CLIA-waived test. (Urine test must have a sensitivity of <25 mlU/mL).

   * NOTE: Persons of female sex assigned at birth and of reproductive potential are defined as having reached menarche and have not been post-menopausal for at least 24 consecutive months (i.e. have had menses within the preceding 24 months), and have not undergone testosterone therapy for gender alignment or surgical sterilization such as hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy. An individual's report is considered acceptable documentation or reproductive status.
9. All participants that are participating in sexual activity that could lead to pregnancy must agree to use contraception throughout the study. At least one of the following must be used throughout the study:

   * Diaphragm or cervical cap with spermicide
   * Intrauterine device (IUD)
   * Hormone-based contraceptive
   * Condoms with or without a spermicide

     * NOTE A: Individuals who are not of reproductive potential are not required to use contraception.
     * NOTE B: Sperm-producing participants should refrain from donating sperm during the treatment period and for at least 90 days after the last dose of study treatment.
10. Ability and willingness of individual or legal guardian/representative to provide informed consent.

Exclusion Criteria:

1. Change in the ART regimen within 12 weeks prior to study entry or intended modification of ART during the study.

   * NOTE: Modifications in the dosage or frequency (i.e. twice a day [bid] to once a day [qd]) of individual antiretroviral (ARV) drugs during the 12 weeks prior to study entry are permitted. In addition, the change in formulation (e.g. from standard formulation to fixed-dose combination) is allowed within 12 weeks prior to study entry. A within class single drug substitution (e.g. switch from atazanavir to darunavir, or tenofovir disoproxil fumarate to tenofovir alafenamide) is allowed within 12 weeks prior to study entry. A switch to any other nucleoside reverse transcriptase inhibitor (NRTI) from abacavir (or vice versa) is not permissible. No other changes in ART within the 12 weeks prior to study entry are permitted.
2. Use of any of the following ARV drugs in current regimen: efavirenz, nevirapine, etravirine, lopinavir/ritonavir, and once-daily dosing of raltegravir (bid dosing of raltegravir is acceptable).
3. Two or more HIV-1 RNA determinations >200 copies/mL within 48 weeks prior to study entry.
4. Any febrile illness (>101°F) within 30 days prior to study entry.
5. Use of drugs with anti-CMV activity within 90 days prior to study entry, with the exception of standard dose valacyclovir and acyclovir. See the protocol for more information.
6. Immunosuppressive or immunomodulatory drug use, with the exception of topical, inhaled, and intranasal corticosteroids within 90 days prior to study entry. See the protocol for more information.
7. Concomitant use of prohibited medications. See the protocol for more information.
8. Persons who are breastfeeding, pregnant or planning to become pregnant during the study.
9. Participating in a study where co-enrollment is not allowed.
10. Receipt of any vaccination within 14 days prior to study entry.
11. Presence on screening ECG or a known history of atrial tachycardia (other than sinus tachycardia). Ventricular tachycardia is also an exclusion criterion.
12. History of cardiomyopathy or congenital heart disease or evidence of advanced conduction system disease including second degree heart block Mobitz type II, third degree heart block, AV dissociation or ECG findings that may be suggestive of predisposition to arrhythmia (i.e. delta wave).
13. Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation.
14. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
15. Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to study entry.
16. Known chronic active hepatitis B virus infection within the last 24 weeks prior to study entry.

    * NOTE: Active is defined as hepatitis B surface antigen (HBsAg) positive and hepatitis B DNA (HBV DNA) positive. Persons with HBV DNA below level of quantification (BLQ) for >24 weeks prior to study entry are eligible.
17. Known chronic active hepatitis C within the last 24 weeks prior to study entry.

    * NOTE: Active is defined as a detectable plasma hepatitis C virus (HCV) RNA level. Persons with HCV RNA BLQ for >24 weeks prior to study entry are eligible.
18. Presence of history of conditions that could account for impaired neuropsychological performance (if present), including head injury with prolonged (>1 hour) loss of consciousness, central nervous system infection (e.g. encephalitis), severe learning disability, psychosis, and/or active drug or alcohol use, or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
19. History of multi-class HIV drug resistance or intolerance, such that in the opinion of the investigator, an alternative fully active antiretroviral regimen cannot be constructed should the participant experience loss of viral suppression on their current regimen during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hunt, MD, Study Chair — University of California, San Francisco, HIV/AIDS CRS; Sara Gianella, MD, Study Chair — University of California, San Diego, AntiViral Research Center CRS
Locations (15):
- United States (15):
  - UCSD Antiviral Research Center CRS (Site 701), San Diego, California
  - UCSF HIV/AIDS CRS (Site 801), San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - Weill Cornell Chelsea CRS (7804), New York, New York
  - Weill Cornell Uptown CRS (7803), New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - University of Washington Positive Research CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism with data be made available?
    * Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://submit.mis.s-3.net/. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.
URL: https://submit.mis.s-3.net/

REFERENCES:
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017 — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from 15 US-based sites during the recruitment period of April 2022 to December 2022.
Period: Overall Study
Arm/Group | Letermovir | No Anti-CMV Treatment
Started | 21 | 23
Completed | 10 | 11
Not Completed | 11 | 12
Not completed — Study Terminated by Sponsor | 8 | 9
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Found to Not Meet Eligibility Criteria After Randomization (Never Started Treatment) | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) Population: All enrolled participants who initiated study treatment and all eligible participants in no treatment arm who have initiation of treatment visit
Groups:
- Total: Total of all reporting groups
Arm/Group | Letermovir | No Anti-CMV Treatment | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [55 to 60] | 58 [52 to 62] | 58 [53 to 61]
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1 | 5 | 6
  50-59 years | 12 | 9 | 21
  60-69 years | 5 | 8 | 13
  70 years and above | 1 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth and Use of Gender-Affirming Hormones: Female not taking testosterone (or do not know) | 5 | 7 | 12
  Sex at Birth and Use of Gender-Affirming Hormones: Male not taking feminizing hormones (or do not know) | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 9 | 13 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Screening CD4+ T-cell Count [Count of Participants; unit: Participants]
  <350 cells/mm^3 | 9 | 9 | 18
  ≥350 cells/mm^3 | 10 | 13 | 23
Weight [Median (Inter-Quartile Range); unit: kg] | 90.9 [70.9 to 99.8] | 87.9 [77.7 to 106.1] | 90.3 [75.8 to 101.0]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.1 [25.0 to 32.8] | 29.4 [25.6 to 31.3] | 29.4 [25.4 to 32.4]
Body Mass Index Category [Count of Participants; unit: Participants]
  Underweight (<18.5) | 1 | 0 | 1
  Normal (18.5-24.9) | 4 | 5 | 9
  Overweight (25-29.9) | 5 | 7 | 12
  Obese (≥30) | 9 | 10 | 19
Antiretroviral Therapy Regimen [Count of Participants; unit: Participants]
  BIC/FTC/TAF | 4 | 7 | 11
  DOR/DTG/FTC/TDF | 0 | 1 | 1
  DTG/3TC | 1 | 2 | 3
  DTG/ABC/3TC | 3 | 2 | 5
  DTG/FTC/TAF | 4 | 2 | 6
  EVG/COBI/FTC/TAF | 4 | 2 | 6
  RPV/CAB | 1 | 2 | 3
  RPV/DRV/COBI/FTC/TAF | 1 | 0 | 1
  RPV/DTG | 1 | 2 | 3
  RPV/DTG/FTC/TAF | 0 | 1 | 1
  RPV/FTC/TAF | 0 | 1 | 1
CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 380 [268 to 809] | 461 [317 to 677] | 384 [281 to 677]
HIV-1 RNA [Count of Participants; unit: Participants] — Participants in the <20, <40, and <128 copies/mL groups had assay results below the limit of quantification.
  Participants
    <20 copies/mL | 11 | 13 | 24
    <40 copies/mL | 5 | 6 | 11
    <128 copies/mL | 1 | 0 | 1
    ≥Lower Limit of Quantification | 2 | 3 | 5
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] — Population: Only quantifiable HIV-1 RNA records were log-transformed, where quantifiable HIV-1 RNA is defined as greater than or equal to the lower limit of quantification
  log10 copies/mL
    number analyzed (Participants) | 2 | 3 | 5
    (all) | 1.49 [1.30 to 1.68] | 1.49 [1.34 to 1.78] | 1.49 [1.34 to 1.68]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 14.2 [13.8 to 15.0] | 14.2 [13.1 to 14.6] | 14.2 [13.6 to 14.8]
Platelet Count [Median (Inter-Quartile Range); unit: platelets/mm^3] | 215000 [180000 to 238000] | 231500 [179000 to 294000] | 215000 [180000 to 272000]
Creatinine Clearance [Median (Inter-Quartile Range); unit: mL/min] | 87.4 [78.1 to 112.3] | 86.8 [75.6 to 109.9] | 87.4 [77.2 to 109.9]
eGFR [Median (Inter-Quartile Range); unit: mL/min/1.73 m^2] — Population: eGFR reporting was optional
  mL/min/1.73 m^2
    number analyzed (Participants) | 14 | 14 | 28
    (all) | 80.0 [66.0 to 87.0] | 75.0 [68.0 to 84.0] | 77.5 [66.5 to 86.5]
Soluble TNF Receptor Type II (sTNFRII) [Mean (Standard Deviation); unit: log10 pg/mL] — Population: Baseline sTNFRII was only calculated for participants in the per-protocol population, where baseline refers to the average of study entry and treatment initiation measures
  log10 pg/mL
    number analyzed (Participants) | 17 | 22 | 39
    (all) | 3.39 (0.12) | 3.40 (0.10) | 3.39 (0.11)
Soluble TNF Receptor Type II [Median (Inter-Quartile Range); unit: log10 pg/mL] — Population: Baseline sTNFRII was only calculated for participants in the per-protocol population, where baseline refers to the average of study entry and treatment initiation measures
  log10 pg/mL
    number analyzed (Participants) | 17 | 22 | 39
    (all) | 3.37 [3.30 to 3.45] | 3.39 [3.34 to 3.45] | 3.39 [3.31 to 3.45]

OUTCOME MEASURES:

1. Primary Outcome: Change (Absolute) in sTNFRII
Description: The absolute change in sTNFRII from Baseline (average of study entry and treatment initiation visits) to Week 46/48 (average of Week 46 and Week 48), or the latest result in the treatment phase. Linear regression was used to estimate the mean change. The covariates were study arm and the gender and CD4 stratification factors.
Time Frame: Measured at Baseline and Weeks 46 and 48
Population: Per-protocol population: All mITT participants who did not prematurely discontinue study product prior to Week 8, had self-reported adherence >50% (letermovir arm only) and did not have a confirmed HIV-1 virologic failure during the treatment phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 pg/mL
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
log10 pg/mL | -0.028 [-0.064 to 0.008] | 0.003 [-0.029 to 0.036]
Statistical Analysis 1: Comparison: Letermovir vs No Anti-CMV Treatment; Test type: Superiority; p = 0.20, Regression, Linear — No adjustment for multiple comparisons; Mean Difference (Net) = -0.031, 95% CI 2-sided [-0.080 to 0.018] — Treatment effect was estimated as the difference in mean change in log10 sTNFRII with randomized letermovir compared to no anti-CMV treatment from a linear regression model (0 reflects no difference between arms)

2. Secondary Outcome: Occurrence of Grade ≥3 AEs or Confirmed HIV-1 Virologic Failure
Description: Adverse events were graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), corrected Version 2.1, July 2017. Adverse events were graded on a scale from 1-5: 1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death.
  Confirmed virologic failure was defined as two consecutive HIV-1 RNA levels ≥200 copies/mL by real-time HIV-1 RNA testing. Participants with a plasma HIV-1 RNA ≥200 copies/mL at any visit had a confirmatory viral load obtained as soon as possible but within 14 days after the first sample was drawn, if possible. If the consecutive measurement of HIV-1 RNA was also ≥200 copies/mL, the participant was considered to have confirmed virologic failure.
Time Frame: Measured from study entry through Week 48
Population: Modified intent to treat population: all eligible, randomized participants excluding letermovir arm participants who did not initiate study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 19 | 22
Participants | 5 | 2
Statistical Analysis 1: Comparison: Letermovir vs No Anti-CMV Treatment; Test type: Superiority; p = 0.19, Chan/Zhang exact test diff. proportions — No adjustment for multiple comparisons; Risk Difference (RD) = 0.172, 95% CI 2-sided [-0.073 to 0.438] — An exact 95% confidence interval around the observed difference in proportions (and the associated p-value) was constructed based on the standardized statistic and inverting two 1-sided tests (Chan-Zhang method)

3. Secondary Outcome: Rate of Change in Odds of Oral CMV DNA Detection
Description: When the number of detection outcomes was sufficient, binary repeated oral CMV DNA detection (yes/no) was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
  Due to the small sample size and small number of detectable CMV DNA results, the GEE model was not able to provide estimates. Cross-sectional CMV DNA detection summaries have been provided instead.
Time Frame: Measured at Baseline and Weeks 8, 46, 48, 52 and 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
Participants
  Baseline: Detected | 2 | 1
  Baseline: Not detected | 15 | 20
  Baseline: No result | 0 | 1
  Week 8: Detected | 0 | 1
  Week 8: Not detected | 15 | 19
  Week 8: No result | 2 | 2
  Week 46: Detected | 0 | 1
  Week 46: Not detected | 12 | 15
  Week 46: No result | 5 | 6
  Week 48: Detected | 0 | 1
  Week 48: Not detected | 13 | 17
  Week 48: No result | 4 | 4
  Week 52: Detected | 0 | 1
  Week 52: Not detected | 12 | 11
  Week 52: No result | 5 | 10
  Week 60: Detected | 0 | 2
  Week 60: Not detected | 8 | 6
  Week 60: No result | 9 | 14

4. Secondary Outcome: Rate of Change in Odds of Genital CMV DNA Detection
Description: When the number of detection outcomes was sufficient, binary repeated genital CMV DNA detection (yes/no) was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
  The model estimates do not reflect the odds of detection, but rather, the change in the odds of detection per week on the multiplicative scale.
Time Frame: Measured at Baseline and Weeks 8, 46, 48, 52 and 60
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: change in odds of detection per week
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
change in odds of detection per week
  Early treatment phase | 0.94 [0.86 to 1.03] | 1.04 [0.96 to 1.13]
  Late treatment phase | 0.95 [0.91 to 0.99] | 1.03 [0.99 to 1.07]
  Post treatment phase | 1.05 [1.01 to 1.09] | 0.89 [0.68 to 1.18]
Statistical Analysis 1: Comparison: Letermovir vs No Anti-CMV Treatment; Early treatment phase comparison; Test type: Superiority; p = 0.12, GEE model for repeated binary outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the early treatment phase; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.80 to 1.03] — Treatment effect was estimated as the odds ratio of weekly rate of change (slope) in odds of CMV DNA detection with randomized letermovir compared to no anti-CMV treatment from a GEE model with linear splines (1 reflects no difference between arms)
Statistical Analysis 2: Comparison: Letermovir vs No Anti-CMV Treatment; Late treatment phase comparison; Test type: Superiority; p = 0.009, GEE model for repeated binary outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the late treatment phase; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.87 to 0.98] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Letermovir vs No Anti-CMV Treatment; Post treatment phase comparison; Test type: Superiority; p = 0.24, GEE model for repeated binary outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the post treatment phase; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.90 to 1.53] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Rate of Change in Odds of Rectal CMV DNA Detection
Description: When the number of detection outcomes was sufficient, binary repeated rectal CMV DNA detection (yes/no) was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
  Due to the small sample size and small number of detectable CMV DNA results, the GEE model was not able to provide estimates. Cross-sectional CMV DNA detection summaries have been provided instead.
Time Frame: Measured at Baseline and Weeks 8, 48 and 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
Participants
  Baseline: Detected | 1 | 1
  Baseline: Not detected | 16 | 21
  Baseline: No result | 0 | 0
  Week 8: Detected | 0 | 0
  Week 8: Not detected | 15 | 20
  Week 8: No result | 2 | 2
  Week 48: Detected | 0 | 2
  Week 48: Not detected | 14 | 15
  Week 48: No result | 3 | 5
  Week 60: Detected | 0 | 0
  Week 60: Not detected | 7 | 8
  Week 60: No result | 10 | 14

6. Secondary Outcome: Rate of Change in Odds of Plasma CMV DNA Detection
Description: When the number of detection outcomes was sufficient, binary repeated plasma CMV DNA detection (yes/no) was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
  Due to the small sample size and small number of detectable CMV DNA results, the GEE model was not able to provide estimates. Cross-sectional CMV DNA detection summaries have been provided instead.
Time Frame: Measured at Baseline and Weeks 8, 46, 48, 52 and 60
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
Participants
  Baseline: Detected | 0 | 0
  Baseline: No detected | 17 | 20
  Baseline: No result | 0 | 2
  Week 8: Detected | 0 | 0
  Week 8: No detected | 16 | 20
  Week 8: No result | 1 | 2
  Week 46: Detected | 0 | 0
  Week 46: No detected | 13 | 16
  Week 46: No result | 4 | 6
  Week 48: Detected | 0 | 0
  Week 48: No detected | 13 | 18
  Week 48: No result | 4 | 4
  Week 52: Detected | 0 | 0
  Week 52: No detected | 11 | 11
  Week 52: No result | 6 | 11
  Week 60: Detected | 0 | 0
  Week 60: No detected | 7 | 8
  Week 60: No result | 10 | 14

7. Secondary Outcome: Rate of Change in sCD163
Description: Repeated, continuous sCD163 was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
Time Frame: Measured at Baseline and Weeks 8, 24, 46, 48, 52 and 60
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 ng/mL/week
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
log10 ng/mL/week
  Early treatment phase | 0.0012 [-0.0031 to 0.0055] | 0.0010 [-0.0038 to 0.0057]
  Late treatment phase | -0.0005 [-0.0012 to 0.0003] | 0.0002 [-0.0007 to 0.0012]
  Post treatment phase | 0.0028 [-0.0001 to 0.0057] | -0.0028 [-0.0083 to 0.0027]
Statistical Analysis 1: Comparison: Letermovir vs No Anti-CMV Treatment; Early treatment phase comparison; Test type: Superiority; p = 0.95, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the early treatment phase; Mean Difference (Net) = 0.0002, 95% CI 2-sided [-0.0062 to 0.0066] — Treatment effect was estimated as the difference in weekly rate of change (slope) in log10 sCD163 with randomized letermovir compared to no anti-CMV treatment from a GEE model with linear splines (1 reflects no difference between treatment groups)
Statistical Analysis 2: Comparison: Letermovir vs No Anti-CMV Treatment; Late treatment phase comparison; Test type: Superiority; p = 0.28, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the late treatment phase; Mean Difference (Net) = -0.0007, 95% CI 2-sided [-0.0019 to 0.0005] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: Letermovir vs No Anti-CMV Treatment; Post treatment phase comparison; Test type: Superiority; p = 0.077, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the post treatment phase; Mean Difference (Net) = 0.0056, 95% CI 2-sided [-0.0006 to 0.0118] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: Rate of Change in sTNFRII
Description: Repeated, continuous sTNFRII was modeled with generalized estimating equations (GEE) to estimate the weekly rate of change (slope). The covariates were study arm and the gender and CD4 stratification factors, as well as a three-level period effect (early treatment phase [through Week 8], late treatment phase, post-treatment phase) and its interaction with the study arm.
Time Frame: Measured at Baseline and Weeks 8, 24, 46, 48, 52 and 60
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 pg/mL/week
Arm/Group | Letermovir | No Anti-CMV Treatment
Number analyzed (Participants) | 17 | 22
log10 pg/mL/week
  Early treatment phase | 0.0009 [-0.0032 to 0.0050] | 0.0000 [-0.0027 to 0.0026]
  Late treatment phase | -0.0010 [-0.0019 to -0.0001] | -0.0001 [-0.0009 to 0.0007]
  Post treatment phase | 0.0001 [-0.0015 to 0.0018] | -0.0021 [-0.0050 to 0.0007]
Statistical Analysis 1: Comparison: Letermovir vs No Anti-CMV Treatment; Early treatment phase comparison; Test type: Superiority; p = 0.72, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the early treatment phase; Mean Difference (Net) = 0.0009, 95% CI 2-sided [-0.0040 to 0.0058] — Treatment effect was estimated as the difference in weekly rate of change (slope) in log10 sTNFRII with randomized letermovir compared to no anti-CMV treatment from a GEE model with linear splines (1 reflects no difference between arms)
Statistical Analysis 2: Comparison: Letermovir vs No Anti-CMV Treatment; Late treatment phase comparison; Test type: Superiority; p = 0.13, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the late treatment phase; Mean Difference (Net) = -0.0009, 95% CI 2-sided [-0.0022 to 0.0003] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 3: Comparison: Letermovir vs No Anti-CMV Treatment; Post treatment phase comparison; Test type: Superiority; p = 0.17, GEE model for repeated outcomes — No adjustment for multiple comparisons; P-value is from the time and treatment group interaction in the post treatment phase; Mean Difference (Net) = 0.0023, 95% CI 2-sided [-0.0010 to 0.0055] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: From study entry to Week 60, or premature study discontinuation
Description: The DAIDS AE Grading Table (Version 2.0) was used for grading adverse events:
  * Grade ≥3 AEs
  * All AEs that led to a change in study treatment/intervention regardless of grade
  * All AEs meeting SAE definition or EAE reporting requirement
  * All Grade ≥2 cardiac arrhythmias (i.e., atrial fibrillation, atrial flutter, etc.)
  * Any Grade ≥1 SARS-CoV-2 or monkeypox infection or AE related to these infections (including any related signs or symptoms Grade ≥1)
  * Any acute febrile illness (>101°F)
Arm/Group | Letermovir | No Anti-CMV Treatment
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/22
Other Adverse Events (participants affected / at risk) | 9/19 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letermovir (N=19) | No Anti-CMV Treatment (N=22)
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Failed back surgery syndrome (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letermovir (N=19) | No Anti-CMV Treatment (N=22)
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 4
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Priapism (Reproductive system and breast disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations include the open-label design and the premature study closure leading to a small sample size and differential time in the treatment phase between the two arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04840199/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT04840199/SAP_001.pdf